CLINICAL TRIAL: NCT05826730
Title: Investigation of The Effect of Eccentric Muscle Training on Pain and Functionality in People With Non-Specific Neck Pain
Brief Title: Eccentric Exercise in Patients With Non-Specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021 / 16
Record Dates: First submitted 2023-02-15; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Neck Pain
Keywords: Neck pain; Exercise; Eccentric strengthening; Pain; Disability
MeSH Terms: conditions — Neck Pain; Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: Randomized-controlled study
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Active Comparator): Eccentric muscle training for neck muscles
  Interventions: Other: Eccentric Exercises
- Control (No Intervention): Home exercise program for neck muscles

INTERVENTIONS:
Other: Eccentric Exercises — Eccentric Exercises for neck muscles.
  Arms: Exercise

SUMMARY:
Neck pain is one of the most frequently investigated and common musculoskeletal disorders that cause disability in the community.If neck pain is due to multifactorial etiology, it is defined as non-specific neck pain.Eccentric exercises are used to increase muscle strength and muscle mass.

Non-specific neck pain affects negatively and often leads to severe disability. Various rehabilitation techniques are available to reduce pain and disability and increase functional level.

This study aimed to compare the pain and functional status of eccentric exercise training and home program exercise groups of people with non-specific neck pain.

DETAILED DESCRIPTION:
It is known that exercise treatments are useful in strengthening neck muscles and controlling postural disorders in patients with neck pain, which is currently accepted. Eccentric exercises are used to increase muscle strength and muscle mass.

Home exercise and eccentric exercise training groups were included in a total of 24 sessions (8 weeks*3 days); home exercise program was applied to the individuals in the control group. Visual Analog Scale, Mc Gill Melzack Pain Assessment, Neck Disability Index, hand grip strength, and skin resistance assessments.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Non-Specific neck pain by a physician
* Having a complaint of non-specific neck pain for at least 3 months
* Neck pain severity >40mm according to VAS
* Voluntary participation of the individual in the study

Exclusion Criteria:

* Radiculopathy and structural defect in the cervical region,
* Surgical history on the cervical region,
* Inflammatory disease,
* Severe psychological illness,
* Presence of infection in bone and soft tissue in the cervical spine,
* Malignancy,
* Advanced osteoporosis,
* Having upper extremity pathologies,
* Having a neurological disease that will prevent treatment
* Having previously undergone cervical region and spine surgery
* To be included in the physiotherapy program from the neck and back region in the last 6 months,
* In case of administration of drugs such as NSAIDs, opioids in the last 24 hours

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Pain Characteristics | before 8 weeks and end of the 8 weeks.
  Pain frequency, duration
Pain severity | before 8 weeks and end of the 8 weeks.
  Visual analog scale-VAS
Mcgill- Melzack Pain Questionnaire | before 8 weeks and end of the 8 weeks.the 24 session.
  Mcgill- Melzack Pain Questionnaire

SECONDARY OUTCOMES:
Disability | before 8 weeks and end of the 8 weeks.
  Neck Disability index
Hand grip strength | before 8 weeks and end of the 8 weeks.
  Digital Hand Dynamometer
Skin resistance | before 8 weeks and end of the 8 weeks.
  Digital Multimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
no sharing of any participant's data